CLINICAL TRIAL: NCT03417076
Title: A Phase 1, Single Center, Open-label, Single Period, Non-randomized Study to Determine the Absolute Bioavailability of Bexagliflozin Tablets Following a Single Oral Dose Co-administered With an Intravenous Microtracer Dose of 14C-Bexagliflozin in Healthy Male Subjects
Brief Title: Absolute Bioavailability Study With Bexagliflozin
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to not initiate study due to sufficient bioavailability information
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THR-1442-C-446
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — bexagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bexagliflozin (Experimental): Each subject will receive a single oral dose of bexagliflozin tablets, 20 mg, followed by a single IV dosing of < 30 ug 14C-bexagliflozin in 0.9% saline solution).
  Interventions: Drug: Bexagliflozin

INTERVENTIONS:
Drug: Bexagliflozin — Bexagliflozin tablets, 20 mg, and bexagliflozin by IV
  Other Names: EGT0001442, EGT0001474

SUMMARY:
The purpose of this study is to determine the absolute bioavailability of bexagliflozin following a single oral dose co-administered with an intravenous dose.

ELIGIBILITY:
Inclusion Criteria:

* body-mass index (BMI) between 18.0 kg/m2 and 32.0 kg/m2
* no nicotine and tobacco consumption in the past 3 months
* willing and able to be confined to the clinical research facility as required by the protocol

Exclusion Criteria:

* clinically significant history of allergy to drugs or latex
* history of alcohol or drug dependence in the past 12 months.
* donation of a significant amount of blood in the past 2 months
* willing to use an adequate form of birth control during the study and for 90 days after discharge from clinic
* exposure to investigational drug in the past 30 days or 7 half-lives of the investigational drug, whichever is longer

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2018-09-16 (Estimated); Study Completion 2018-09-16 (Estimated)

PRIMARY OUTCOMES:
absolute bioavailability (Fp.o.) of bexagliflozin tablets | Up to 48 hours
  oral to IV ratio of dose-normalized AUC0-inf (area under the plasma concentration time curve extrapolated to infinity)

SECONDARY OUTCOMES:
adverse events | Up to 3 days
  adverse event as a measure of safety and tolerability of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mason Freeman, M.D., Study Director — Massachusetts General Hospital
Locations (1):
- Clinical Research Site, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No